CLINICAL TRIAL: NCT05169580
Title: A Phase 1 Open-Label, Multiple-Dose Study to Evaluate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of FTX-6058 in Subjects With Sickle Cell Disease (SCD)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Pociredir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6058-SCD-101
Record Dates: First submitted 2021-12-14; First posted 2021-12-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Pharmacokinetics; Pharmacodynamics; Pociredir; Open label
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Open-label, multiple-dose study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pociredir oral capsule(s) in Sickle Cell participants (Experimental): Cohort 1 will receive 6 mg of Pociredir by mouth once daily. Cohort 2 will be dosed at 2 mg once daily by mouth, and cohort 3 will be dosed at 12 mg once daily by mouth. The Sponsor will reinitiate enrolment in the 3rd cohort (12 mg cohort) with the updated inclusion and exclusion criteria. Based on review of available safety and biomarker data and with the recommendation of the DMC, a subsequent 4th cohort of 20 mg and potentially a 5th cohort of 30 mg may be initiated. A total of seven cohorts may be included. Following the first cohort, doses for all subsequent cohorts will be determined following DMC review of the safety and pharmacokinetic data observed in participants from the prior and ongoing cohorts. Alternate dosing schedules may be evaluated in some of the cohorts.
  Interventions: Drug: Pociredir oral capsule(s)

INTERVENTIONS:
Drug: Pociredir oral capsule(s) — Participants will receive Pociredir
  Other Names: FTX-6058

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of Pociredir in participants with sickle cell disease.

DETAILED DESCRIPTION:
This is a Phase 1 multicenter, international, open-label study evaluating the safety, tolerability, pharmacokinetics (PK), fetal hemoglobin (HbF) induction and biological activity of Pociredir in participants 18-65 years of age, inclusive, with SCD.

Participants will receive 12 weeks of dosing with 4 weeks of follow-up. Approximately 10 participants will be enrolled in each cohort. A maximum of 3 participants with SCD HbSC+ genotype may be enrolled in each cohort.

Cohort 1 will receive 6 milligrams (mg) of Pociredir by mouth once daily. Doses for subsequent cohorts will be determined following review by the Data Monitoring Committee [DMC]. A total of seven cohorts may be included. Cohort 2 will be dosed at 2 mg once daily by mouth, and cohort 3 will be dosed at 12 mg once daily by mouth. The Sponsor will reinitiate enrolment in the 3rd cohort (12 mg cohort) with the updated inclusion and exclusion criteria. Based on review of available safety and biomarker data and with the recommendation of the DMC, a subsequent 4th cohort of 20 mg and potentially a 5th cohort of 30 mg may be initiated. Additional cohorts using alternative dosing schedules may be considered based on available data.

The primary endpoints of the study are to evaluate the safety and tolerability of Pociredir as measured by the frequency of adverse events and to evaluate single and multiple-dose pharmacokinetics of Pociredir in participants with sickle cell disease. Secondary endpoints include evaluating the effect of Pociredir on fetal hemoglobin induction in peripheral blood and evaluating the effects of Pociredir on hemolysis in participants with sickle cell disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is 18 to 65 years of age, inclusive at the time informed consent is obtained.
* Documented SCD at the time of screening (S/S, S/β0, S/β+, and S/C only) as confirmed through review of medical records or HPLC.
* Participants who meet at least one the following criteria:

  1. ≥4 to 10 episodes of SCD pain crisis over 12 months, or ≥2 to 5 over 6 months prior to screening
  2. ≥2 episodes of SCD pain crisis plus at least one of the following over previous 12 months: i) Acute chest syndrome (ACS) ii. Hepatic or splenic sequestration iii. Priapism
  3. ≥2 of the following events over the previous 12 months:i. ACS ii. Hepatic or splenic sequestration iii. Priapism
  4. Tricuspid regurgitant jet velocity (TRV) ≥ 3.0 meter/second(m/s) OR TRV ≥ 2.5 m/s + N-terminal pro b-type natriuretic peptide (NT-proBNP) plasma level ≥ 160 picogram per milliliter; OR documented ongoing pulmonary hypertension diagnosed from previous echocardiogram or right-sided heart catheterization with mean pulmonary artery pressure > 25 millimeter of mercury;
  5. SCD-related chronic kidney disease (CKD)
  6. Meet medical criteria to receive (e.g., post-cerebrovascular accident) but are contraindicated for chronic transfusions (e.g., alloimmunization, transfusion reactions)
* Previous experience with Hydroxyurea (HU) but have shown to be unresponsive and/or intolerant or ineligible AND
* Previous experience with a stable dose of voxelotor, crizanlizumab, and/ or L-glutamine but have shown to be unresponsive and/or intolerant or ineligible
* Per Investigator's recommendation, participants may continue crizanlizumab and/or L-glutamine but must be on a stable dose for at least 6 months
* HbF ≤ 20% of total Hb
* Total Hb ≥ 5.5 g/dL and ≤ 12 g/dl (males) or ≤ 10.6 g/dl (females) at screening.
* Participant must meet both of the following laboratory values at screening:

  1. Absolute neutrophil count ≥ 1.5 × 10^9 per liter (/l)
  2. Platelets ≥ 80 × 10^9/l
  3. Absolute reticulocyte count at screening ≥ 100 x 10^9/l.

Key Exclusion Criteria:

* Sickle cell complication requiring care from a medical provider in hospital or emergency care setting in the 14 days prior to starting study drug.
* History of bone marrow transplant or human stem cell transplant or gene therapies.
* • Participants with a history of severe renal disease defined as estimated glomerular filtration rate < 30 mL/min/1.73m^2. Participants on dialysis of any kind are excluded.
* Participants receiving regularly scheduled transfusions or therapeutic phlebotomies, or any participant who has been transfused within 60 days prior to initiating study drug.
* Participant with active malignancy, or history of cancer (except for squamous cell skin cancer, basal cell skin cancer, and stage 0 cervical carcinoma in situ, with no recurrence for the last 5 years), or has an immediate family member with known or suspected familial cancer syndrome. Known presence of a chromosomal abnormality or genetic mutation that may put the participant at an increased risk of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Participant currently on HU, or have received HU, within 60 days prior to initiating study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | Up to approximately 16 weeks of monitoring
  To evaluate the safety and tolerability of Pociredir in adult participants with sickle cell disease based on the frequency of adverse events (AEs) and changes in clinically significant laboratory test results, vital signs and electrocardiograms (ECGs) parameters.
Plasma Concentrations of Pociredir | Days 1, 14, 28, 42, 56, 70, 84 and 91
  Blood samples will be collected to measure the plasma concentration of Pociredir at specified timepoints.

SECONDARY OUTCOMES:
Change from Baseline in percentage fetal hemoglobin (%HbF) biomarkers in peripheral blood | Baseline and at Days 1, 14, 28, 42, 56, 70, 84, 91, and 112
  The percentage of HbF will be measured in peripheral whole blood.
Change from Baseline in % Reticulocytes | Baseline and at Days 1, 14, 28, 42, 56, 70, 84, 91, and 112
  The percentage of reticulocytes will be measured in peripheral whole blood.
Change from Baseline in Absolute Reticulocyte Count | Baseline and at Days 1, 14, 28, 42, 56, 70, 84, 91, and 112
  The absolute reticulocyte count will be measured in peripheral whole blood.
Change from Baseline in Red cell distribution width | Baseline and at Days 1, 14, 28, 42, 56, 70, 84 and 91
  Blood samples will be collected for the analysis of hematology parameter: red cell distribution width
Change from Baseline in unconjugated bilirubin | Baseline and at Days 1, 14, 28, 42, 56, 70, 84 and 91
  Blood samples will be collected for the analysis of clinical chemistry parameter: unconjugated bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Adeyemi Adenola, MD, Study Director — Fulcrum Therapeutics
Locations (18):
- United States (14):
  - University of Arkansas for Medical Sciences (UAMS), Little Rock, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - Sonar Research Center, Atlanta, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Queens Hospital Cancer Center, Jamaica, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Eastern Carolina University, Greenville, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - University of Texas Houston, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Nigeria (3):
  - National Hospital, Abuja, Abuja
  - University of Ibadan, Ibadan
  - Barau Dikko Teaching Hospital, Kaduna
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, South Africa

REFERENCES:
- [Background] Ngo DA, Aygun B, Akinsheye I, Hankins JS, Bhan I, Luo HY, Steinberg MH, Chui DH. Fetal haemoglobin levels and haematological characteristics of compound heterozygotes for haemoglobin S and deletional hereditary persistence of fetal haemoglobin. Br J Haematol. 2012 Jan;156(2):259-64. doi: 10.1111/j.1365-2141.2011.08916.x. Epub 2011 Oct 24. PMID 22017641
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290
- [Background] Sankaran VG, Orkin SH. The switch from fetal to adult hemoglobin. Cold Spring Harb Perspect Med. 2013 Jan 1;3(1):a011643. doi: 10.1101/cshperspect.a011643. PMID 23209159
- [Background] Saraf SL, Molokie RE, Nouraie M, Sable CA, Luchtman-Jones L, Ensing GJ, Campbell AD, Rana SR, Niu XM, Machado RF, Gladwin MT, Gordeuk VR. Differences in the clinical and genotypic presentation of sickle cell disease around the world. Paediatr Respir Rev. 2014 Mar;15(1):4-12. doi: 10.1016/j.prrv.2013.11.003. Epub 2013 Nov 15. PMID 24361300
- [Background] Steinberg MH, Chui DH, Dover GJ, Sebastiani P, Alsultan A. Fetal hemoglobin in sickle cell anemia: a glass half full? Blood. 2014 Jan 23;123(4):481-5. doi: 10.1182/blood-2013-09-528067. Epub 2013 Nov 12. PMID 24222332
- [Derived] Abbasi M, Srivastava A, Saraf SL. Management of Kidney Disease with Sickle Cell Disease. J Am Soc Nephrol. 2025 Oct 1;36(10):2041-2054. doi: 10.1681/ASN.0000000804. Epub 2025 Jun 26. PMID 40569673